CLINICAL TRIAL: NCT00674388
Title: The Pediatric Anesthesia Quality Improvement Project
Acronym: WUS
Status: Recruiting | Type: Observational
Sponsor: The Society for Pediatric Anesthesia (Other)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other); Monroe Carell Jr. Children's Hospital at Vanderbilt (Other); Seattle Children's Hospital (Other); Boston Children's Hospital (Other); Emory-Children's Center (Other); Baylor College of Medicine (Other); Johns Hopkins University (Other); Children's Hospital Los Angeles (Other); Morgan Stanley Children's Hospital (Other); Children's Hospital of Philadelphia (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other); University of Pittsburgh (Other); Phoenix Children's Hospital (Other); University of Michigan (Other); Children's National Health System, Washington DC (Unknown); Arkansas Children's Hospital Research Institute (Other); Children's Hospital Colorado (Other); St. Jude Children's Research Hospital (Other); Cook Children's Health Care System (Other); SSM Cardinal Glennon Children's Medical Center (Unknown); The Children's Hospital at Montefiore (Other); Children's Medical Center Dallas (Other); Lucile Packard Children's Hospital Stanford (Unknown); Alfred I. duPont Hospital for Children (Other); Johns Hopkins All Children's Hospital (Other); Children's Hospitals and Clinics of Minnesota (Other); Oakland Medical Center (Other); Children's Hospital and Medical Center, Omaha, Nebraska (Other); Medical University of South Carolina (Other); Akron Children's Hospital (Other); Women & Children's Hospital of Buffalo (Other); Dayton Children's Hospital (Other); Riley Children's Hospital (Unknown); Cleveland Clinic Children's Hospital (Unknown); Dell Children's Medical Center of Central Texas (Other); Le Bonheur Children's Hospital (Other); Arnold Palmer Hospital for Children (Other); University of Iowa (Other); Shriners Hospitals for Children (Other); Penn State Hershey Children's Hospital (Unknown)
Responsible Party: Principal Investigator, Jayant K Deshpande, MD MPH, Executive Director, Wake up Safe, The Society for Pediatric Anesthesia
Other Study IDs: Wake up Safe
Record Dates: First submitted 2008-05-05; First posted 2008-05-07 (Estimated); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Surgery; Anesthesia; Children
Keywords: Children; Anesthesia; Surgery; Complication

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No

SUMMARY:
The Study is designed to collect information about adverse events that occur in children undergoing anesthesia in participating hospitals. Demographic information will be collected on all anesthetics. An analysis of each adverse event will be performed and entered into the database. From this information we will devise strategies to prevent these adverse events.

ELIGIBILITY:
Inclusion Criteria:

* All children undergoing anesthesia at participating hospitals

Exclusion Criteria:

* Patients over 21 years of age

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All Children undergoing anesthesia at the participating hospitals
Sampling Method: Non-Probability Sample
Enrollment: 5000000 (Estimated)
Dates: Start 2008-02 (Actual); Primary Completion 2035-12 (Estimated); Study Completion 2040-12 (Estimated)

PRIMARY OUTCOMES:
number of adverse events | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jayant K Deshpande, MD MPH, MD, Study Director — The Society for Pediatric Anesthesia
Locations (37):
- United States (37):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital Los Angeles, Los Angeles, California
  - Oakland Medical Center, Oakland, California
  - Lucile Packard Children's Hospital Stanford, Palo Alto, California
  - Colorado Children's Hospital, Aurora, Colorado
  - Nemours/Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Health System, Washington D.C., District of Columbia
  - Arnold Palmer Children's Hospital, Orlando, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Emory Children's Center, Atlanta, Georgia
  - Children's Memorial Hospital, Chicago, Illinois
  - University of Iowa Stead Family Children's Hospital, Iowa City, Iowa
  - Johns Hopkins Childrens Center, Baltimore, Maryland
  - Children's Hospital Boston, Boston, Massachusetts
  - University of Michigan CS Mott Children's Hospital, Ann Arbor, Michigan
  - SSM Cardinal Glennon Health Care System, St Louis, Missouri
  - Children's Hospital and Medical Center, Omaha, Nebraska
  - Womens and Childrens Hospital of Buffalo, Buffalo, New York
  - Morgan Stanley Children's Hospital, New York, New York
  - Children's Hospital at Montefiore, New York, New York
  - Akron Children's Hospital, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Children's Hospital, Cleveland, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - Penn State Hershey Children's Hospital, Hershey, Pennsylvania
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Pittsburgh Children's Hospital, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - LeBonheur Children's Hospital, Memphis, Tennessee
  - St Jude Children's Research Hospital, Memphis, Tennessee
  - Monroe Carell Jr Children's Hospital at Venderbilt, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Children's Medical Center Dallas, Dallas, Texas
  - Cook Children's Health Care System, Fort Worth, Texas
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington